CLINICAL TRIAL: NCT02014857
Title: Evaluation of GCF MMP-1, -8 and Growth Factor Levels in Smokers With Periodontal Health
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gülnihal Eren, Research Asisstant, Research Assistant, Ege University
Other Study IDs: Ege University
Record Dates: First submitted 2013-12-10; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Smoking, Healthy Volenteers
Keywords: Smoking, gingival crevicular fluid, matrix metalloproteinases, intercellular signaling peptides and proteins, healthy volunteers
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Periodonatlly healthy smokers: Gingival crevicular fluid sampling
  Interventions: Procedure: Gingival Crevicular Fluid Sampling
- Periodontally healhty non-smokers: Gingival crevicular fluid sampling
  Interventions: Procedure: Gingival Crevicular Fluid Sampling

INTERVENTIONS:
Procedure: Gingival Crevicular Fluid Sampling

SUMMARY:
Increased levels of cytokines in GCF have been demonstrated in smoker subjects with chronic periodontitis. It is not surprising that increased levels of inflammation associated molecules in GCF has been observed in smokers with periodontitis. However, it is not clear if smoking has an influence on these parameters in periodontally healthy individuals. In the present study, it has been hypothesized that smoking might affect the levels of GCF MMPs and growth factors in young adults with periodontal health.

DETAILED DESCRIPTION:
The main objective of the present study was to investigate the GCF levels of MMP-1, MMP-8, TGF-β1, PDGF-AB and VEGF in smoker versus non-smoker periodontally healthy young adults.

A total of 32 periodontally healthy young adults including 16 smokers and 16 non-smokers, were recruited for the present cross-sectional study ( 18 female and 14 males; age range: 19 to 27 years).

All participants had a thorough full-mouth clinical examination. The measurement of probing depth (PD) and clinical attachment level (CAL) were assessed at six sites per tooth in the whole mouth, excluding third molars in all study participants. Bleeding on probing (BOP) and the amount of plaque accumulation were also evaluated.

GCF sampling sites were selected from the sites without BOP and plaque accumulation. GCF samples were obtained from buccal aspects of proximal sites in a single-rooted teeth in each individual participating in the present study. Paper strips† were carefully inserted 1 mm into the crevice for 30 seconds. Care was taken to avoid mechanical trauma. The absorbed GCF volume was estimated by a calibrated instrument. Then each strip from each patient were placed into one polypropylene tube before freezing at -40°C. The readings were converted to an actual volume (µl) reference to the standard curve. All GCF samples were stored at -40°C until the laboratory analyses.

Considering a difference of 50% in mean GCF levels of the biochemical markers and assuming standard deviations to be maximum 80% of the mean values and accepting a power of 90%, P value of 5% in smoker and non-smoker groups, minimum sample size was calculated.

Chi-square test was used to determine for differences in gender and smoking state between the study groups. Student t test was applied for comparison of age between smokers and non-smokers. Normality test was performed to evaluate the distribution of clinical periodontal parameters and levels of growth factor and MMP-1, -8. Growth factor and MMP levels were compared by Mann-Whitney U test in study groups.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally and systemically healthy individuals
* Have at least 20 teeth
* >10 cigarettes/day consumption for smoker group
* Non-smokers subjects were selected from periodontally healthy participants who had never smoked.

Exclusion Criteria:

* Any health condition affecting their systemic status such as diabetes mellitus, immunologic disorders, human immunodeficiency virus infections, hepatitis were excluded
* Also pregnant and lactating women and those taking oral contraceptive drugs were not included in the study.
* Any antibiotic intake within the last 3 months and any periodontal treatment within 6 months

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental faculty students
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
GCF levels of MMP-1, MMP-8, TGF-β1, VEGF and PDGF-AB | Baseline
  Total amount and concentration of these biomarkers in GCF

CONTACTS AND LOCATIONS:
Overall Officials: Gul Atilla, Professor, Study Director — Ege University School of Dentistry; Hatice Oya Turkoglu, Assoc. Professor, Study Chair — Ege University School of Dentistry; Harika Atmaca, PhD, Study Chair — Celal Bayar University
Locations (1):
- Ege University School of Dentistry Department of Periodontology, Izmir, Turkey (Türkiye)